CLINICAL TRIAL: NCT07370727
Title: Effects of Velocity-Based Resistance Training on Renal Function and Metabolic Health in Kidney Transplant Recipients: Protocol for a Randomized Controlled Trial
Brief Title: Velocity-Based Resistance Training in Kidney Transplant Recipients
Acronym: VBRTKIDNEY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universitaria del Area Andina (Other)
Responsible Party: Principal Investigator, Jhonatan Camilo Peña Ibagon, Principal Investigator, PhD Candidate in Sport and Exercise Science and Technology", Fundación Universitaria del Area Andina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CV2025-IMED-B-13434
Record Dates: First submitted 2025-09-30; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant Recipients; Metabolic Syndrome; Cardiovascular Risk Factors
Keywords: Kidney Transplant; Renal Transplant; Velocity based resistance training; Metabolic Health; Exercise Intervention; Glomerular Filtration Rate (eGFR)
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Maximal Velocity Group (Experimental): Participants will perform velocity-based resistance training at maximal intended concentric velocity. Training load will progress from 20% to 60% of 1RM. Each set will be terminated once a 20% loss of movement velocity is reached.
  Interventions: Other: Velocity-Based Resistance Training - Maximal Velocity Protocol
- Submaximal Velocity Group (Active Comparator): Participants will perform supervised velocity-based resistance training for 12 weeks, 3 sessions per week. Each repetition will be executed at approximately 50% of maximal concentric velocity. Training load will progress from 20% to 60% of 1RM, with sets completed according to a predetermined number of repetitions (20-30 depending on load).
  Interventions: Other: Velocity-Based Resistance Training - Submaximal Velocity Protocol

INTERVENTIONS:
Other: Velocity-Based Resistance Training - Submaximal Velocity Protocol — A 12-week supervised resistance training program performed 3 sessions per week. Exercises will include bench press, squat, and shoulder press in Smith machine. Participants will execute each repetition at ~50% of maximal concentric velocity, with sets completed according to predetermined repetitions (20-30 depending on load, 20-60% 1RM).
  Arms: Submaximal Velocity Group
Other: Velocity-Based Resistance Training - Maximal Velocity Protocol — A 12-week supervised resistance training program performed 3 sessions per week. Exercises will include bench press, squat, and shoulder press in Smith machine. Participants will execute each repetition at maximal concentric velocity, with sets terminated at 20% velocity loss. Training loads will increase progressively (20-60% 1RM).
  Arms: Experimental - Maximal Velocity Group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of velocity-based resistance training on renal function and metabolic health in kidney transplant recipients. Participants will be randomized into two groups performing resistance training at different execution velocities (maximal intended vs. submaximal controlled). The intervention will last 12 weeks and include multi-joint exercises (squat, bench press, military press). Primary outcomes include renal function (serum creatinine, eGFR, blood urea nitrogen, uric acid) and metabolic markers (HDL, triglycerides, glucose, waist circumference, blood pressure). Secondary outcomes include muscle strength, force-velocity profile, anthropometry, physical activity, fitness perception, and adherence to immunosuppressive medication.

DETAILED DESCRIPTION:
This randomized controlled trial will examine the physiological and metabolic responses to different resistance training velocities in kidney transplant recipients. Participants will be randomized to perform either maximal-velocity or submaximal-velocity resistance exercises for 12 weeks. Each session will include multi-joint movements (bench press, squat, overhead press) using a Smith machine. Training loads will be individualized (20-60% 1RM) and monitored using a linear encoder to control velocity loss. Primary endpoints are renal function and metabolic health markers, while secondary outcomes include neuromuscular performance and adherence to immunosuppressive therapy. The study has received ethics approval from Fundación Universitaria del Área Andina (Acta 15, April 22, 2025).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 50 years.
* Kidney transplant performed ≥12 months before enrollment.
* Stable graft function in the previous 6 months (serum creatinine < 1.5 mg/dL, no rejection episodes).
* Written medical clearance from a nephrologist to perform moderate-to-vigorous physical activity.
* Signed informed consent.

Exclusion Criteria:

* Active autoimmune disorders.
* Recent coronary disease (≤6 months).
* Severe musculoskeletal limitations incompatible with resistance training.
* Diagnosis of diabetes mellitus (pre- or post-transplant).
* Current active infection.
* Use of immunosuppressive drugs with contraindications for exercise (e.g., mTOR inhibitors at baseline).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine (mg/dL) - change from baseline | Baseline and week 13 (after completion of 12-week intervention)
  Serum creatinine will be measured from venous blood samples processed in an external certified laboratory (IDIME, Bogotá). This parameter will serve as a biomarker of renal graft function.
Estimated glomerular filtration rate (eGFR, mL/min/1.73 m²) - change from baseline | Baseline and week 13 (after completion of 12-week intervention)
  The estimated glomerular filtration rate (eGFR) will be calculated from serum creatinine using validated equations (CKD-EPI or MDRD). This measure will serve as the most sensitive indicator of renal graft function.
Blood urea nitrogen (BUN, mg/dL) - change from baseline | Baseline and week 13 (after completion of 12-week intervention)
  Blood urea nitrogen will be measured to monitor renal clearance capacity and metabolic status.
Serum Uric Acid (mg/dL) | Baseline and week 13 (after completion of 12-week intervention)
  Serum uric acid will be measured as a biomarker of renal excretory capacity and cardiovascular risk.
HDL cholesterol (mg/dL) - change from baseline | Baseline and week 13 (after completion of 12-week intervention)
  HDL cholesterol will be measured as a protective lipid biomarker inversely associated with metabolic and cardiovascular risk.
Triglycerides (mg/dL) - change from baseline | Baseline and week 13 (after completion of 12-week intervention)
  Serum triglycerides will be measured to evaluate metabolic health and risk of cardiovascular disease.
Fasting glucose (mg/dL) - change from baseline | Baseline and week 13 (after completion of 12-week intervention)
  Fasting blood glucose will be measured through enzymatic methods to evaluate glycemic control.
Waist circumference (cm) - change from baseline | Baseline and week 13 (after completion of 12-week intervention)
  Waist circumference will be measured at the narrowest point of the torso, midway between the lower margin of the ribs and the iliac crest, following ISAK recommendations. This anthropometric variable will serve as a key component of metabolic syndrome diagnosis.
Metabolic Risk Index (z-score composite) | Baseline and week 13 (after completion of 12-week intervention)
  A composite metabolic risk index will be calculated from triglycerides, LDL, HDL, glucose, and systolic/diastolic blood pressure values. Each variable will be standardized as z-scores; HDL will be multiplied by -1 due to its inverse relationship with cardiovascular risk. The final score will be the sum of standardized values.

SECONDARY OUTCOMES:
Handgrip strength | Baseline and week 13 (after completion of 12-week intervention)
  Handgrip strength will be assessed using a digital dynamometer (Takei Scientific Instruments, Tokyo). Two trials per hand, best value recorded. This test reflects overall muscle strength.
Body Composition (fat percent, muscle percent, visceral fat) | Baseline and week 13 (after completion of 12-week intervention)
  Body composition will be assessed using segmental bioelectrical impedance analysis (Tanita IRONMAN BC-1500). Measurements will include fat percentage, muscle percentage, and visceral fat.
Force-Velocity Profile | Baseline and week 13 (after completion of 12-week intervention)
  :The force-velocity profile will be assessed using a linear encoder (T-Force) during three multi-joint exercises (bench press, squat, overhead press). The relationship between force and velocity will be calculated to estimate neuromuscular performance.
Body Height (cm) | Baseline and week 13 (after completion of 12-week intervention)
  Body height will be measured with a digital stadiometer following the Frankfurt plane reference to ensure standardized posture.
Relative Handgrip Strength (kg/kg body weight) | Baseline and week 13 (after completion of 12-week intervention)
  Relative handgrip strength will be calculated by dividing the maximum handgrip force by body weight to account for body size.
Comorbidity and Immunosuppressive Therapy Questionnaire | Baseline and week 13 (after completion of 12-week intervention)
  A structured questionnaire will be used to record comorbidities and medication adherence. Adherence will be rated on a 5-point Likert scale (1 = never adherent, 5 = always adherent), where higher scores indicate better adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Colombia, Bogotá, Bogota D.C., Colombia

REFERENCES:
- [Background] Michou V, Nikodimopoulou M, Liakopoulos V, Anifanti M, Papagianni A, Zembekakis P, Deligiannis A, Kouidi E. Home-Based Exercise Training and Cardiac Autonomic Neuropathy in Kidney Transplant Recipients with Type-II Diabetes Mellitus. Life (Basel). 2023 Jun 14;13(6):1394. doi: 10.3390/life13061394. PMID 37374177
- [Background] Pena JC, Sanchez-Guette L, Lombo C, Pinto E, Collazos C, Tovar B, Bonilla DA, Cardozo LA, Tellez LA. Characterization of Load Components in Resistance Training Programs for Kidney Transplant Recipients: A Scoping Review. Sports (Basel). 2025 May 19;13(5):153. doi: 10.3390/sports13050153. PMID 40423289
- [Background] Lima PS, de Campos AS, de Faria Neto O, Ferreira TCA, Amorim CEN, Stone WJ, Prestes J, Garcia AMC, Urtado CB. Effects of Combined Resistance Plus Aerobic Training on Body Composition, Muscle Strength, Aerobic Capacity, and Renal Function in Kidney Transplantation Subjects. J Strength Cond Res. 2021 Nov 1;35(11):3243-3250. doi: 10.1519/JSC.0000000000003274. PMID 31714457
- [Background] Hernandez Sanchez S, Carrero JJ, Morales JS, Ruiz JR. Effects of a resistance training program in kidney transplant recipients: A randomized controlled trial. Scand J Med Sci Sports. 2021 Feb;31(2):473-479. doi: 10.1111/sms.13853. Epub 2020 Oct 23. PMID 33038051
- See also: Fundación Universitaria del Área Andina — https://www.areandina.edu.co